CLINICAL TRIAL: NCT01810666
Title: Routine Prophylaxis Treatment Versus On-demand Treatment for Children With Severe Hemophilia A: Comparison of All Bleeding Events in Chinese Hemophilia Patients
Brief Title: Prophylaxis Versus on Demand Treatment for Children With Hemophilia A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16287; 2014-001362-10 (EudraCT Number)
Record Dates: First submitted 2013-03-12; First posted 2013-03-13 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recombinant Factor VIII (Experimental)
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Participants received Recombinant Factor VIII (Rec. factor VIII) on-demand treatment for 12 weeks followed by a 12 weeks prophylaxis treatment phase. The dose and mode of prophylaxis treatment was 25 IU/Kg, 3 times/per week. The dose in on-demand treatment was decided by physician according to the package insert or the current standard of care.

SUMMARY:
Comparison of the effect of three times a week prophylaxis on all bleeds with on-demand treatment for children with severe Hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 2-16yrs
* Severe hemophilia A (<1% FVIII:C [Blood Clotting Factor VIII:C] )
* Minimum of at least 50 documented ED (exposure day) prior to enrolment
* No measurable inhibitor activity at baseline and history of FVIII inhibitor antibody formation
* Parents or legal guardians document, sign, and date informed consent

Exclusion Criteria:

* Another bleeding disease that is different from hemophilia A
* Known hypersensitivity to the active substance, mouse or hamster protein
* Thrombocytopenia (platelet count <100 000/mm3) based on previous medical records

Ages: 2 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- China (4):
  - Guangzhou, Guangdong
  - Wuhan, Hubei
  - Beijing
  - Tianjin

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment period was between 20-Mar-2013 to 28-Jun-2013.
Pre-assignment Details: Of 33 participants who were screened for inclusion in the study, 30 were enrolled and received treatment.
Groups:
- Rec. Factor VIII On-demand Followed by Prophylaxis: Participants received Recombinant Factor VIII (Rec. factor VIII) on-demand treatment for 12 weeks followed by a 12 weeks prophylaxis treatment phase. The dose and mode of prophylaxis treatment was 25 IU/Kg, 3 times/per week. The dose in on-demand treatment was decided by physician according to the package insert or the current standard of care.
Period: Overall Study
Arm/Group | Rec. Factor VIII On-demand Followed by Prophylaxis
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rec. Factor VIII On-demand Followed by Prophylaxis
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 30
  Others | 0
Baseline weight [Mean (Standard Deviation); unit: Kg] | 41.42 (19.02)
Baseline body mass index [Mean (Standard Deviation); unit: Kg/m2] | 18.65 (4.16)
Target Joint for Bleeds [Number; unit: Participants]
  No | 8
  Yes | 22
Number of Target Joint [Number; unit: Participants]
  0 | 8
  1 | 16
  2 | 6
Prior FVIII Treatment On-demand [Number; unit: Participants] | 30
Number of Bleeds in Last 3 Months [Mean (Standard Deviation); unit: Bleeds] | 12.4 (8.71)
Number of Joint Bleeds in Last 3 Months [Mean (Standard Deviation); unit: Bleeds] | 8.73 (8.07)

OUTCOME MEASURES:

1. Primary Outcome: Difference of Annualized Number of All Bleeds Between On-demand and Prophylaxis Period
Description: Annualized bleedings period 1 minus period 2 ITT analysis set.
Time Frame: Week 1-12 (on-demand treatment) and 13-24 (prophylactic treatment)
Measure: Median (95% Confidence Interval); unit: Bleeds
Arm/Group | Rec. Factor VIII On-demand Followed by Prophylaxis
Number analyzed (Participants) | 30
Bleeds | 56.00 [48.80 to 62.54]

2. Secondary Outcome: Difference of Annualized Number of Joint Bleeds Between On-demand and Prophylaxis Period
Description: Annualized joint bleedings period 1 minus period 2 ITT analysis set.
Time Frame: Week 1-12 (on-demand treatment) and 13-24 (prophylactic treatment)
Measure: Median (95% Confidence Interval); unit: Bleeds
Arm/Group | Rec. Factor VIII On-demand Followed by Prophylaxis
Number analyzed (Participants) | 30
Bleeds | 37.71 [30.42 to 46.02]

3. Secondary Outcome: Difference of Intra-individual Change of Joint Function During Each Period Assessed by the Hemophilia Joint Health Score Between On-demand and Prophylaxis Period
Description: Hemophilia Joint Health Score(HJHS) ranges from 0 to 124. Higher values in the HJHS represent worse situation for the subject. 2-sided Hodges Lehmann estimates for median 95% CI HJHS values difference of changes ITT analysis set.
Time Frame: From baseline to Week 12 (on-demand treatment) and Week 24 (prophylactic treatment)
Measure: Median (95% Confidence Interval); unit: Scores on scale
Arm/Group | Rec. Factor VIII On-demand Followed by Prophylaxis
Number analyzed (Participants) | 30
Scores on scale | -3.00 [-5.00 to 0.00]

ADVERSE EVENTS:
Time Frame: From first treatment through 3 days after the last dose of study drug, up to 6 months
Arm/Group | Rec. Factor VIII On-demand Followed by Prophylaxis
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rec. Factor VIII On-demand Followed by Prophylaxis (N=30)
Pyrexia (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days